CLINICAL TRIAL: NCT05849948
Title: The Effect of Chronobiological Nutritional Approach on Growth and Breastfeeding Processes of Premature Babies
Brief Title: Effect Of Chronobıologıcal Nutrıtıon On Premature Babıes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ezgi Ayvaz, NURSE, Eskisehir Osmangazi University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: YENİDOĞAN DOKTORA TEZ
Record Dates: First submitted 2023-04-18; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Nutrition, Healthy
Keywords: premature; chorobiological nutrition; Breastfeeding Processes
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- choronobiological nutrition group (Experimental): newborns were fed according to chronobiological nutrition
  Interventions: Behavioral: choronobiological nutrition
- control group (No Intervention): newborns will be fed in the order in which breastmilk is delivered to the hospital

INTERVENTIONS:
Behavioral: choronobiological nutrition — Providing infant nutrition in accordance with crinobiological nutrition
  Arms: choronobiological nutrition group

SUMMARY:
The aim of this study is to determine the effect of chronobiological nutrition approach on the growth and breastfeeding processes of premature babies. It will be carried out in a randomized controlled experimental design. In the study, it is planned to have 2 groups as experimental and control. As a result of the power analysis using the G Power 3.0.10 program, 90% power; A total of at least 78 samples were found to be sufficient in the study with a 5% margin of error (n1: 39; n2: 39). However, considering that the case could be lost, it was decided to increase it by 20% to 94 babies. Infants will be assigned to groups using a stratified sequential block randomization method. Premature babies will be stratified by week of gestation, birth weight and sex, and then an equal number of babies will be assigned to each group by blocking.

The appointment of premature infants will be decided by sequential block randomization.

After the descriptive information of the babies assigned to the groups is recorded in the questionnaire, the experimental group will be fed by applying the chronobiological nutrition approach. The control group will be fed without applying the chronobiological nutrition approach. The discharge times will be calculated for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Being treated in the NICU
* Gestation week is between 30 and 36
* The delivery took place in the hospital where the study was conducted.
* 70% of the daily enteral feeding is done with breast milk

Exclusion Criteria:

* The baby is less than 30 weeks of gestation and greater than 36 weeks of gestation.
* Having neurological sequelae
* Having Grade 4 intraventricular bleeding
* The development of problems such as sepsis, NEC, which may change the general condition
* Being followed in invasive mechanical ventilation
* Receiving narcotic analgesics and sedation
* The baby has been shipped from outside
* Having undergone gastrointestinal (GIS) surgery or having GIS anomaly

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The change in the discharge time of newborns will be evaluated by using a questionnaire prepared by the researcher. | The newborn will be evaluated once a week for up to an average of 6 weeks after the date of hospitalization.
  newborn was evaluated during hospital treatment

SECONDARY OUTCOMES:
Weight gain of newborns will be evaluated using a questionnaire prepared by the investigator. | The newborn will be evaluated once a week for up to an average of 6 weeks after the date of hospitalization.
  newborn was evaluated during hospital treatment

OTHER OUTCOMES:
Height growth of newborns will be evaluated using a questionnaire prepared by the researcher. | The newborn will be evaluated once a week for up to an average of 6 weeks after the date of hospitalization.
  newborn was evaluated during hospital treatment
Head circumference of newborns will be evaluated using a questionnaire prepared by the researcher. | The newborn will be evaluated once a week for up to an average of 6 weeks after the date of hospitalization.
  newborn was evaluated during hospital treatment
The duration of breastfeeding of newborns by their mothers will be evaluated using a questionnaire prepared by the researcher. | will be evaluated once a month for 6 months after discharge
  The newborn was evaluated in the first 6 months after discharge.